CLINICAL TRIAL: NCT07119814
Title: Comparison of Outcome of Safe T Separators and Conventional Elastomeric Separators
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber College of dentistry (Other)
Responsible Party: Principal Investigator, Haris Mustafa, Dr., Khyber College of dentistry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59/RRB/KCD
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group A was assigned to Conventional elastomeric separators and group B to safe T separator group (Other): Placement of conventional elastomeric separators and safe T separators intraorally in patients coming for fixed orthodontic treatment.
  Interventions: Device: Conventional Separators placement; Device: Safe T separator

INTERVENTIONS:
Device: Conventional Separators placement — Safe T separators and conventional elastomeric separators will be placed in patients of fixed orthodontic treatment.
Device: Safe T separator — Safe T separators will be placed in patients of fixed orthodontic treatment

SUMMARY:
All participants in this study will be provided with information concerning the study's objectives, and benefits associated with participation. Participants will be informed that their involvement in this study presents no potential risks associated with their participation. Written consent will be obtained with appropriate information provided. Demographic data like age, BMI, gender, residence, socio economic status, occupation status, and literacy status will be documented. Patients undergoing fixed orthodontic treatment will be allocated in two groups equally by using the blocked randomization technique. Patients in Group A will undergo safe-T separators i.e initial thickness of Safe-T separators will be 1mm, Patients in Group B will undergo conventional elastomeric separators i.e thickness of elastomeric separators will be 1.2 mm. Separators will be positioned on either side of lower arch, each type of separator will be in sites, resulting in a sites within the lower arch. A separator placement tool will be utilised to position the separators. The comprehensive assessment will be carried out under the supervision of a consultant possessing at least five years of post-fellowship experience. Patient data will be recorded using a predefined structured proforma.

ELIGIBILITY:
Inclusion Criteria:

* Age range (18-40) Years Male/Female Patients undergoing fixed orthodontic treatment as mentioned in operational

Exclusion Criteria:

* Patients with poor oral hygiene Patients with periodontal conditions Patients failed to provide consent form

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Amount of Pain | Pain will be measured over 3 days of stsrting treatment
  Measuring the amount of pain caused by the two modalities of treatment using visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber college of dentistry peshawar, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No